CLINICAL TRIAL: NCT01948791
Title: 16 Weeks Interventional Study on Titration and Dose/Efficacy Assessment of Exelon (Rivastigmine) in Chinese Alzheimer's Disease Patients (INSTINCT)
Brief Title: 16w Interventional Study on Titration and Dose/Efficacy Assessment of Exelon in Chinese Alzheimer's Disease Patients
Acronym: INSTINCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713BCN05
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; ENA713; Chinese patients; INSTINCT
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENA713 (Experimental): Patients had a dose escalation from 3mg/d to 12mg/d to reach individual tolerated dosage during the titration period of 12 weeks.
  Interventions: Drug: ENA713

INTERVENTIONS:
Drug: ENA713 — The following strengths of Rivastigmine capsules were provided: Rivastigmine capsule strengths: 1.5mg, 3mg, 4.5mg. The 6mg dose was administered as one 1.5mg capsule and one 4.5mg capsule, and when necessary, the 3mg dose could also be administered as two 1.5mg capsules. Rivastigmine was administered from 3mg/d at baseline. Then dose escalation was made in 3mg/d increments, at a minimun of 4 weeks between dose increases to a maximum dose of 12mg/d or the individual's best tolerated dose.
  Other Names: Rivastigmine

SUMMARY:
To investigate the efficacy of Exelon capsule at maximal tolerated dose in mild to moderate Chinese AD patients via dosage titration from 3mg/d to 12mg/d in a 16 weeks duration

ELIGIBILITY:
Key Inclusion Criteria:

* Have a diagnosis of dementia of the Alzheimer's type according to the DSM-IV criteria and have a clinical diagnosis of probable AD according to NINCDS/ADRDA criteria
* MMSE score of ≥ 10 and ≤ 26
* The treatment naïve patient and the one who have stopped the donepezil, galantamine, huperzine A, or memantine at least 2 weeks
* Be in stable medical condition
* Have signed off informed consent form by patients or his/her legal guardian

Key Exclusion Criteria:

* Severe AD
* Patients with a history of cerebrovascular disease, Active or uncontrolled epilepsy, Active hypothyroidism, asthma, CNS infection, other Neurodegenerative disorders, an advanced, severe, progressive, or unstable medical condition
* Attending other clinical trials or taking other clinical trial drugs
* A score of > 4 on the Modified Hachinski Ischemic Scale (MHIS);
* Patients who is using any AChEI or memantine

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, MD/PhD, Principal Investigator — Department of Neurology, Xuanwu HospitalCapital Medical University, Beijing, P.R.China
Locations (1):
- Novartis Investigative Site, Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 222 patients were screened/enrolled to this study but 41 did not receive study drug.
Pre-assignment Details: The Intention analysis set consists of 165 patients who received at least 1 treatment & had at least 1 assessment on primary efficacy variables.
Period: Overall Study
Arm/Group | ENA713
Started | 222
Completed | 151
Not Completed | 71
Not completed — Adverse Event | 12
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 6
Not completed — Management issues | 1
Not completed — Others | 7
Not completed — Screening failure | 35

BASELINE CHARACTERISTICS:
Population: Subjects who received at least one treatment, and had at least one post-baseline assessment on primary efficacy variables.
Arm/Group | ENA713
Number analyzed (Participants) | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (8.4)
Gender [Count of Participants; unit: Participants]
  Female | 101
  Male | 64

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog)
Description: The Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) was used to measure change in cognitive function. Alzheimer's disease assessment scale (ADAS) is a scale to measure specific cognitive and behavior disorders in Alzheimer disease (AD) patients. The Alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog) provides a total score range 0-70, and consists of 11 items with lower score indicating lighter impairment and higher total scores indicating more impairment. A negative change score indicates improvement from baseline. Two-sided 95% CI of the difference in the means between baseline and post-baseline values were calculated.
Time Frame: Baseline, Week 16
Population: The Per Protocol (PP) population included all patients who had been enrolled to receive treatment, and who had received at least 1 dose of study drug, had 1 baseline assessment & at least 1 post-baseline efficacy assessment for primary efficacy variable within the Week 16 visit window, and had no major protocol violations.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ENA713
Number analyzed (Participants) | 151
units on a scale | -2.0 [-3.0 to 1.1]
Statistical Analysis 1: Comparison: ENA713; The hypothesis to test the non-inferiority of post-baseline change in ADAS-Cog from baseline was: H0: μP - μB ≥ 1.40, Ha: μP - μB < 1.40 where μP and μB are the ADAS-Cog score (actual) at 16 weeks of Rivastigmine treatment and the baseline ADAS-Cog score (actual), respectively; Test type: Non-Inferiority or Equivalence — If the upper limit of the 95% confidence interval of the mean difference between the baseline score and post-baseline score falls on the left of MeanP-MeanB+1.40, the post-baseline noninferiority to baseline can be concluded. If the upper limit of the 95% confidence interval of the mean difference between the baseline score and post-baseline score falls on the left of 0, superiority can be concluded; p < 0.001, t-test, 1 sided

2. Secondary Outcome: Change From Baseline in the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Score
Description: ADCS-ADL is a scale based on caregiver's assessment of patient's activities of daily life. It is used in clinical studies on dementia & consists of 23 items and is designed to assess patient's basic & instrumental activities of daily life, such as the abilities necessary for personal care, communicating & interacting with other people, maintaining a household, conducting hobbies & interests, & making judgments & decisions. Response to each item is obtained by interview with the caregiver. The basic activities of daily life domain includes mandatory options for best response, or "yes" or "no" questions with separate sub-questions. Higher score & more "yes" answers indicate better level of self-care of patient. Therefore the higher the total score is, the better the patient's functions. The total score is the sum of the scores of all the items & sub-questions,& ranges from 0 to 78. Two-sided 95% CI of the difference in the means between baseline and post-baseline values were calculated.
Time Frame: Baseline, Week 16
Population: The Per Protocol (PP) population included all patients who had been enrolled to receive treatment, had received at least 1 dose of study drug, had 1 baseline assessment & at least 1 post-baseline efficacy assessment for primary efficacy variable within the Week 16 visit window & had no major protocol violations.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ENA713
Number analyzed (Participants) | 151
units on a scale | 0.9 [-0.5 to 2.3]

3. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE)
Description: MMSE was used to determine patient's eligibility to participate, is an easy & practical screening test to identify cognitive disorders. Test consists of 2 parts: language (time orientation, registration & attention) & performance (recall, response to written/verbal commands, writing ability & reproduction of complex polygons); total score range: 0-30; higher score = better function. Positive change score = improvement from baseline. To meet eligibility criteria, patient's MMSE total score at screening had to be 10-26 (inclusive). Interpretation of MMSE by 4 methods: Single Cut0ff: <24=abnormal; Range: <21=Increased odds of dementia; >25=Decreased odds of dementia; Education: 21- abnormal for 8th grade education, <23=abnormal for high school education, <24=abnormal for college education; Severity: 24-30=no cognitive impairment, 18-23=mild cognitive impairment, 0-17=severe cognitive impairment. 2-sided 95% CI of difference in means between baseline & post-baseline values were calculated
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ENA713
Number analyzed (Participants) | 151
units on a scale | 0.3 [-0.4 to 0.8]

4. Secondary Outcome: Mean Change From Baseline in Neuropsychiatric Inventory (NPI) Score
Description: This scale assesses a larger scope of the behavior problems/disorders experienced in dementia patients, and identifies the frequency & severity of the behavior disorders, & allows rapid assessment using screening questions. 10 questions in behavior domain & 2 in autonomic nervous system domain were assessed by the investigator interviewing with the caregiver. The NPI-12 total score is the total score of the 12 items, among which the score for each domain is the product of frequency (range: 1-4 points) and severity (range: 1-3 points). The highest score for each domain is 12 points and all the domains have the same weight. Therefore the range of NPI-12 total score is 0-144 points. The NPI-10 total score is the total score of the first 10 items 0-120, which constitute the original form of this scale. A higher NPI total score indicates more severe behavior disorder. Two-sided 95% CI of the difference in the means between baseline and post-baseline values were calculated.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ENA713
Number analyzed (Participants) | 151
units on a scale
  NPI-10 | -3.6 [-5.3 to -1.9]
  NPI-12 | -4.0 [-6.2 to -1.9]

5. Secondary Outcome: Change From Baseline in Caregiver Burden Inventory (CBI) Score
Description: CBI, formulated by Novak and Guest in 1989, is a relatively complete and effective scale to measure caregiver burden that has been extensively adopted internationally. CBI has a total of 24 items in 5 domains, i.e., time dependency items (items 1-5), development items (items 6-10), physical health items (items 11-14), social relations items (items 15-18), and emotional heath items (items 19-24). Each item is scored on a 5-point scale based on the intensity of burden (0-4 points), so that the total score is 0-96, a higher score indicating heavier burden. It is a self-administered scale that takes about 10-15 minutes to complete. Two-sided 95% CI of the difference in the means between baseline and post-baseline values were calculated.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ENA713
Number analyzed (Participants) | 151
units on a scale | -1.4 [-3.1 to 0.4]

ADVERSE EVENTS:
Description: The safety set consists of 181 patients who received at least one drug treatment and had post-baseline safety assessments.
Arm/Group | ENA713
Serious Adverse Events (participants affected / at risk) | 7/181
Other Adverse Events (participants affected / at risk) | 69/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENA713 (N=181)
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Pneumocephalus (Injury, poisoning and procedural complications) | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Brain injury (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ENA713 (N=181)
Abdominal discomfort (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 37
Vomiting (Gastrointestinal disorders) | 30
Decreased appetite (Metabolism and nutrition disorders) | 14
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 6

LIMITATIONS AND CAVEATS:
Of the total recruited subjects, 181 subjects received at least one drug treatment and there were post-baseline safety assessment. They were incorporated into the safety population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data in the clinical trial.